CLINICAL TRIAL: NCT04289935
Title: Intelligent Vacuum Assisted Biopsy Immediately Before Surgery As an Intra- or Pre-Operative Surrogate for Patient Response to Neoadjuvant Chemotherapy for Breast Cancer (VISION I): a Multicenter Prospective Feasibility Trial
Brief Title: Intelligent Vacuum Assisted Biopsy Immediately Before Surgery As an Intra- or Pre-Operative Surrogate for Patient Response to Neoadjuvant Chemotherapy for Breast Cancer
Acronym: VISION I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Hirslanden, Zurich (Other)
Collaborators: Oncoplastic Breast Consortium (OPBC) (Unknown)
Responsible Party: Principal Investigator, PD Dr. med. Christoph Tausch, Principal Investigator, Klinik Hirslanden, Zurich
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HIRSLANDEN 01 OPBC SAKK 23/18
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; VISION I; breast cancer; Vacuum assisted biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, single arm, feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): * Unicentric histologically confirmed invasive luminal B, HER2- enriched, triple negative breast cancer + Clipping + Neoadjuvant chemotherapy
  * rCR / near-rCR in MRI / US
  * Registration
  * US-guided VAB
  * Breast conserving surgery / mastectomy
  * Pathology examination 1. Preoperative VAB, 2. Surgical specimen
  Interventions: Procedure: Vacuum assisted biopsy (VAB)

INTERVENTIONS:
Procedure: Vacuum assisted biopsy (VAB) — The trial intervention consists of a diagnostic interventional procedure, US-guided or mammographically guided VAB post-NAC, prior to the standard breast surgery.

SUMMARY:
Neoadjuvant chemotherapy (NAC) is common practice in the primary treatment of breast cancer, leading to a complete pathologic remission (pCR) of the tumor in more than 50% in aggressive tumor types. As NAC induces different response patterns, radiologic imaging is not sufficiently accurate in predicting residual disease. Because of this uncertainty, surgery is so far the only valid option to either ascertain complete response or to remove the complete residual disease.

Vacuum-assisted biopsy (VAB) with the possibility of obtaining tissue of the former tumor center could contribute more reliably to detect any residual tumor or respectively, rule out residual disease. Ultrasound (US) or mammographically (MG) guided VAB will be used in this trial in order to detect residual tumor lesions in patients with radiological complete response (rCR) after NAC. The investigators will evaluate the diagnostic accuracy of the post-NAC VAB sample in comparison to the sample obtained in open surgery.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NAC), initially indicated to downstage tumors to achieve the option of breast conserving surgery, has lately become common practice in the primary treatment of breast cancer. The use of modern NAC regimens lead to a complete pathologic remission (pCR) of the tumor in more than 50% in aggressive tumor types.

In general, it is difficult to predict pCR in the absence of invasive surgical techniques, as it depends on several factors such as biological subtype, the used chemotherapy regimen and anatomic stage. The most common imaging methods beside clinical examination are breast ultrasound, mammography and breast magnetic resonance imaging (MRI). As NAC induces different response patterns, radiologic imaging is not sufficiently accurate in predicting residual disease. Because of this uncertainty, surgery (and the standardized assessment of resected tissue) is so far the only valid option to either ascertain complete response or to remove the complete residual disease.

Vacuum-assisted biopsy (VAB) with the possibility of obtaining tissue of the former tumor center could contribute more reliably to detect any residual tumor or respectively, rule out residual disease. Ultrasound (US) or mammographically (MG) guided VAB will be used in this trial in order to detect residual tumor lesions in patients with radiological complete response (rCR) after NAC. The investigators will evaluate the diagnostic accuracy of the post-NAC VAB sample in comparison to the sample obtained in open surgery.

The main objective of the trial is to determine the diagnostic accuracy of I-VAB using the full pathologic specimen evalutation obtained after open surgery to detect residual tissue.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* unifocal, histologically confirmed invasive breast cancer with IHC luminal B (with or without overexpression or amplification of the HER2 receptor) and all ER negative (ER < 10%) breast cancers
* Initial tumor size larger than 1 and less than 5 cm (cT1c to cT2), any N, M0
* Clipping of the primary tumor center prior to the start of neo-adjuvant chemotherapy
* Neo-adjuvant chemotherapy resulting in a radiological complete response or near complete response on MR-Imaging (confirmed within 28 days before or on registration) as described in the trial specific MR-Imaging instructions (available on the welcome page of the study specific SecuTrial link). MRI is strongly recommended, alternative ultrasound
* Former tumor bed must be accessible for biopsy
* Female or male aged ≥ 18 years
* Adequate condition for breast cancer surgery
* Patients with a previously treated malignancy are eligible, when the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low

Exclusion criteria:

* Metastatic breast cancer
* Multifocal/Multicentric breast cancer
* Inflammatory breast cancer
* Luminal-A types of breast cancers (ER ≥ 10% and PgR ≥ 10 % and G1 or 2, and/or Ki-67 ≤ 20%, HER2 negative) or low risk if assessed by a validated genomic prognostic test (e.g. Mammaprint, Endopredict, Oncotype or Nanostring)
* Distinct radiological sign of residual disease in the breast after neo-adjuvant chemotherapy by imaging
* Intra-/peritumoral microcalcifications larger than 2 cm at time of diagnosis
* Any local therapy (irradiation or surgery) to the currently treated breast prior to the trial intervention
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, trial intervention and follow-up, affect patient compliance or place the patient at high risk from trial intervention-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | max. 6 weeks after registration
  Sensitivity of I-VAB is defined as proportion of true positive patients (Both VAB and surgery showing non pCR) given patients with non pCR assessed using surgical specimen.

SECONDARY OUTCOMES:
Specificity | max. 6 weeks after registration
  Specificity of I-VAB is defined as proportion of true negative patients (Both VAB and surgery showing pCR) given patients with pCR assessed using surgical specimen.
Positive predictive value (PPV) | max. 6 weeks after registration
  PPV of I-VAB is defined as proportion of true positive patients given patients with non pCR assessed using VAB
Negative predictive value (NPV) | max. 6 weeks after registration
  NPV of I-VAB is defined as proportion of true negative patients given patients with pCR assessed using VAB
Accuracy (ACC) | max. 6 weeks after registration
  ACC of I-VAB is defined as the proportion of true positive and true negative patients.
Surgical lymph node status | max. 6 weeks after registration
  Surgical lymph node status (positive vs. negative) is categorized by the pathologist according to surgical specimen.
Adverse events | From US-guided VAB (max. 6 weeks after registration) until 2 weeks after breast surgery (max 1 day after VAB).
  Proportion of patients with bleeding/hematoma causing immediate surgical intervention and breast infection, which are related to VAB.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Tausch, MD, Study Chair — Brust-Zentrum, Zürich
Locations (26):
- Austria (3):
  - Universitätsspital Salzburg, Salzburg
  - Brustzentrum Schwaz, Schwaz
  - St. Josef Krankenhaus Wien, Vienna
- Germany (4):
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Brustzentrum Heidelberg, Heidelberg
  - UFK Klinikum Südstadt Rostock, Rostock
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Switzerland (18):
  - Tumor Zentrum Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Bethesda Spital, Basel
  - St. Claraspital, Basel
  - Hirslanden Brustzentrum Bern Biel, Bern
  - Kantonsspital Graubünden, Chur
  - Spital Thurgau AG Frauenfeld und Münsterlingen, Frauenfeld
  - Clinique de Genolier, Genolier
  - Luzerner Kantonsspital, Lucerne
  - Hirslanden Klinik St. Anna, Lucerne
  - Ente Ospedaliero Cantonale, Dipartimento di ginecologia e ostretricia, Lugano
  - Brustzentrum Rheinfelden, Rheinfelden
  - Kantonsspital St. Gallen, Sankt Gallen
  - Tumor- und BrustZentrum Ostschweiz, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Brust-Zentrum Seefeld, Zurich
  - Universitäts Spital Zürich, Zurich
- Mediclinic City Hospital Dubai, Dubai, United Arab Emirates